CLINICAL TRIAL: NCT05517187
Title: Clinical Success of Regenerative Endodontic Treatment With Platelets Rich Fibrin PRF as a Secondary Treatment of Mature Necrotic Incisors With Periapical Radiolucency in Adolescents: A Preliminary Parallel Randomized Controlled Clinical Trial
Brief Title: Efficacy of Regenerative Endodontic Treatment With PRF as a Secondary Treatment of Mature Necrotic Incisors in Adolescents
Acronym: PRF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nahda University (Other)
Responsible Party: Principal Investigator, Yassmine mohamed farouk el makawi, Lecturer in pediatric dentistry(clinical investigator), Nahda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 284
Record Dates: First submitted 2022-08-08; First posted 2022-08-26 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Dental Pulp Necroses
Keywords: platelet rich fibrin
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Clot BC (Control arm) (Placebo Comparator): Regenerative endodontic treatment with induced Blood Clot in root canal space as a secondary treatment for failed root canal treated incisors
  Interventions: Other: no intervention
- Platelets Rich Fibrin PRF (Intervention) (Experimental): Regenerative endodontic treatment with Platelet- rich fibrin in root canal space as a secondary treatment for failed root canal treated incisors
  Interventions: Biological: Platelet rich fibrin

INTERVENTIONS:
Other: no intervention — Regenerative endodontic treatment induced with blood clot in root canal space as a secondary treatment for failed root canal treated incisors
  Arms: Blood Clot BC (Control arm)
Biological: Platelet rich fibrin — Regenerative endodontic treatment with platelet rich fibrin in root canal space as a secondary treatment for failed root canal treated incisors
  Arms: Platelets Rich Fibrin PRF (Intervention)

SUMMARY:
Evalaution of clinical success of secondary treatment for total 40 permanent incisors with failed root canal treatment with apical radiolucency.

Twenty of of these permanent incisors will be treated with regenerative endodontic treatment(RET) with platelets rich fibrin PRF as intervention group vs. 20 incisors control group secondary treated with (RET) with induced blood clot (BC).

DETAILED DESCRIPTION:
A preliminary randomized parallel controlled trial will be conducted. Forty teeth of 36 patients were randomly assigned into two groups: group "PRF", treated with RET with PRF platelets rich fibrin (intervention), and group "BC", treated with RET with induced blood clot(control). Upon clinical examination, the presence of pain on biting or percussion, swelling or sinus tract, or abnormal tooth mobility will be considered a failure. To monitor the changes in periapical radiolucency, a periapical index (PAI) will be used. The primary outcome of the current study will be to assess the effectiveness of RET using PRF platelets rich fibrin of mature permanent incisors with periapical radiolucency compared to RET using induced BC formation in the root canal space.

Eligibility criteria:

Healthy adolescents below the age of 18 years who need endodontic retreatment of previously obturated mature single-rooted incisors with gutta-percha will be recruited.

Patients with a positive history of allergic reactions, systemic diseases, and severe emotional or behavioral problems will be precluded. Only teeth diagnosed with asymptomatic apical periodontitis or chronic apical abscess (i.e. little discomfort with intermittent episodes of pus discharge through the sinus tract) were included. To confirm the clinical status, only teeth with a periapical index (PAI) score ≥3 based on Ørstavik et al classification were considered. Teeth with previous attempts for endodontic retreatment including pulpotomy or pulpectomy, non-restorable crowns or need post placement, or periodontal problems were excluded. A tooth must not be a candidate for endodontic surgery according to Glickman et al. indications and the updates of the European Society of Endodontology (e.g. obtaining biopsy, removal of intracanal broken files, persistent periapical lesions standing for a long period, radicular perforation, root fracture, or obstructed root canals, or the inability of complete removal of old gutta-percha or extruded material beyond the apex with persistent apical lesion for long duration).

Interventions:

According to the latest RET operating guidelines issued by the American Academy of Endodontics (AAE) and the European Society of Endodontics (ESE), the standardised operating procedure of RET requires two treatment visits. During the first appointment, infection is controlled and inflammation is relieved with complete removal of failed obturation material. Pulp regeneration and revascularization is accomplished during the second appointment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy patients below age of 18 years.
2. Need endodontic retreatment of previously obturated closed apexes single-rooted incisors with gutta-percha.
3. No previous attempts for endodontic retreatment.
4. Presence of clinical signs and symptoms of chronic apical periodontitis

Exclusion Criteria:

1. Patients with a positive history of allergic reactions, systemic diseases, and severe emotional or behavioral problems were precluded.
2. Teeth with previous attempts for endodontic retreatment including pulpotomy or pulpectomy, non-restorable crowns

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 12 months
  Clinical assessment will be performed at the baseline (T0) and after 12 months (T1). Upon examination, clinical failure will be encountered if one of the following features will present: (i) pain on biting or percussion, (ii) swelling or sinus tract, or (iii) abnormal tooth mobility.
Radiographic success | 12 months
  For a standardized appraisal of the changes in the size of periapical radiolucency, long cone "paralleling technique" with a receptor holder was used after mounting a size II periapical film (Kodak International) to a silicone bite stent.

SECONDARY OUTCOMES:
Pulp sensibility test | 12 months
  In the control and intervention groups, the pulp sensations will be tested with an electric pulp tester (EPT) (Pulp Tester DY 310, Denjoy Dental Co.) at T1 and T2.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Nahda University, Banī Suwayf
  - Nahda, Cairo